CLINICAL TRIAL: NCT03745209
Title: Ultrasound-guided Peripheral IV vs. Standard Technique in Difficult Vascular Access Patients by ICU Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Collaborators: Kingston Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Mohammed Alshamsi, Clinical fellow, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6023923
Record Dates: First submitted 2018-09-09; First posted 2018-11-19 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Difficult IV Access
Keywords: Peripheral IV; Difficult; Ultrasound-guided
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided peripheral IV. (Experimental): Ultrasound-guided peripheral IV cannulation
  Interventions: Device: Ultrasound
- Traditional landmark technique (No Intervention): Traditional landmark technique

INTERVENTIONS:
Device: Ultrasound — Use of real-time ultrasound in an attempt to establish intravenous peripheral catheter.
  Arms: Ultrasound-guided peripheral IV.

SUMMARY:
This is a randomized controlled single-center study that will be conducted in the intensive care unit. The main objective of this study is to assess the success rate of ultrasound-guided peripheral intravenous cannulation in ICU patients with difficult intravenous access compared with traditional landmark technique.

DETAILED DESCRIPTION:
Peripheral IV access is common and essential procedure conducted by nurses in intensive care departments. This important procedure is frequently difficult because of the high prevalence of peripheral edema and obesity among ICU patients. In this study, the investigators will assess the success rate of real-time ultrasound guidance in cannulating difficult access ICU patients. This is a randomized controlled single-site trial with two groups in a parallel design. In this study, the investigators will compare the success rate of ultrasound-guided peripheral intravenous access (experimental group) to a traditional landmark approach (control group) in patients with difficult IV access. It is a non-blinded study because of the nature of the intervention. This study will be conducted in the adult intensive care unit of Kingston general hospital which is an urban university teaching hospital with 33 ICU beds and more than 1000 ICU admissions per year. A sample of ICU patients with difficult cannulation will be selected and enrolled in this study. Difficult cannulation is defined as poorly visible and poorly palpable upper extremities veins due to any cause after two failed attempts using the traditional technique. All consecutive patient with difficult cannulation will be assessed for enrolment in this study starting from October 2018 till March 2019. A research assistant will be available for patient enrollment and data collection between 8:00 AM to 5:00 PM during regular working hours.

The study will be conducted in two phases. Phase 1 will involve education and training of a cohort of nurses to perform US-guided cannulation. Experienced ICU nurses with two years of experience will be recruited to participate in the study. All nurses will have no prior experience in ultrasound-guided peripheral I.V insertion prior to this study. Education consists of didactic 2 hours lecture and hands-on practice on synthetic training models ( blue phantoms). This will cover basic machine operation, image optimization, sonographic anatomy and ultrasound techniques for guiding peripheral I.V cannulation. This will be followed by 2-3 months observation period during which nurses have to perform at least 15 successful ultrasound-guided peripheral cannulations on live subjects before actual patients' enrolment. Phase 2 will involve enrolment of difficult peripheral access ICU patients meeting specific inclusion and exclusion criteria. Patients will be systematically randomized to the ultrasound-guided or the landmark technique using envelop randomization.

Only upper limb veins will be selected for cannulation. All the cannulation will be done under semi aseptic technique as per standard placement and cleaning procedures for peripheral IV access. Ultrasound-guided cannulation will be performed using sterile gel for the procedure and the ultrasound probe will be covered with sterile adhesive films (e.g., 3M Tegaderm). Two already available departmental ultrasound machines (sonosite edge) will be used for this study. High-frequency probe (5-10 MHz) with single operator out of plane (short access) approach will be used for ultrasound-guided cannulation. When using ultrasound for I.V placement, veins deeper than 1.5 cm from the skin surface and veins with a diameter of less than 0.3 cm will be avoided because of high failure rate and increased risk of extravasation. Catheter length and size will be selected based on the depth and size of the veins to ensure that a sufficient portion of the catheter will remain in the vessel to prevent early failure.

Intensive care nurses participating in the study will record all the data related to outcome measures on a preprinted data collection forms.The Investigators will enter the raw data into SPSS software for analysis. An intention-to-treat analysis will be performed. Using the power of 80% and alpha of 0.05, the sample size was calculated to be 25 per group. Categorical variables such as success rate, catheter survival rate and complication rate will be presented as a percentage and will be compared using Fisher exact tests. Continuous variables such as insertion time and the number of attempts will be shown as mean, median (with interquartile ranges), and 95% confidence interval (CI) and will be compared using Mann-Whitney U tests. All statistical analysis will be conducted using IBM SPSS Base 25 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Difficult IV access patients after 2 failed attempts

Exclusion Criteria:

* Upper-extremity cellulitis
* Unstable and need urgent intravenous access( central line or IO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-06-21 (Estimated); Study Completion 2019-06-21 (Estimated)

PRIMARY OUTCOMES:
Overall success rate of IV placement | Up to 30 minutes
  Ability to establish a functioning peripheral IV catheter

SECONDARY OUTCOMES:
Number of skin punctures attempted. | Up to 30 minutes
  An attempt is defined as puncturing skin without need for reinsertion.
24 hours catheter survival | 24 hours post IV insertion
  Functioning catheter 24 hours post insertion
Complications | Up to 7 days
  One of the following is defined as a complication related to peripheral IV insertion: cellulitis, phlebitis, arterial puncture, nerve injuries, infiltration.
  hematoma formation)
Subsequent need for PICC or central line. | Up to 14 days
  Subsequent need for PICC or central line

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed R Alshamsi, MD, Principal Investigator — Kingston Health Sciences Centre
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736

DOCUMENTS (1):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03745209/Prot_000.pdf